CLINICAL TRIAL: NCT03306030
Title: Comparison of Two Split-dose Regimes for Bowel Preparation in Patients With Constipation
Brief Title: Comparison of Two Methods for Bowel Preparation in Patients With Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20172055-2
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Health Behavior
Keywords: PEG; Bowel preparation; Colonoscopy; split-does
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split group (Active Comparator): Split-dose of 4l PEG was used before and on the day of colonoscopy
  Interventions: Drug: Split dose of 4L PEG
- Three times group (Experimental): Three times-dose of 4l PEG was used before and on the day of colonoscop of 4l PEG was used before and on the day of colonoscopy
  Interventions: Drug: Three times dose of 4L PEG

INTERVENTIONS:
Drug: Split dose of 4L PEG — All patients were given oral instruction for bowel preparation on the day of appointment and re-instruction through phone call on two days before scheduled colonoscopy. They were instructed to have a regular lunch and take only clear liquid or low-residual food for the dinner on the day before colonoscopy. The participants began to drink the first 2 L of PEG at 7:00-9 PM on the day before colonoscopy at a rate of 250 mL every 15 minutes. On the day of the procedure, patients took the remaining 2 L 4-6 hours before colonoscopy.
  Arms: Split group
Drug: Three times dose of 4L PEG — The same as mentioned above. The participants began to drink the first 1.5 L of PEG at 2:00 PM and the second 1.5L of PEG at 8:00PM on the day before colonoscopy at a rate of 250 mL every 15 minutes. On the day of the procedure, patients take the remaining 1.0 L 4-6 hours before colonoscopy.
  Arms: Three times group

SUMMARY:
Constipation is a common high risk factor for inadequate bowel preparation. The bowel cleansing efficacy of the standard split-does of 4L seems to be suboptimal in constipated patients. The investigator hypothesized that compared with the standard preparation regime, the split-dose with three times of 4L PEG may be superior in BP quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 with constipation.

Exclusion Criteria:

* History of colorectal surgery BMI>30 Suspected colonic stricture or bowel obstruction Use of purgatives within 3 days Pregnancy or lactation Unable to give informed consent Haemodynamically unstable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of adequate bowel preparation | 1 year
  Adequacy of bowel preparation quality was defined as a total score ≥6 and each segmental score ≥2. The total scores included 3 scores of colonic regions: the right side, the transverse section, and the left side, which ranged from 0 to 9 (0= very poor, 9=excellent). For the unreached colon in incomplete colonoscopy, the segmental BBPS was scored as 0. The total and segmental scores were judged through videos by investigators who were familiar with the criteria and blinded to group allocation.

SECONDARY OUTCOMES:
Adverse event rate | 1 year
Cecal intubation rate | 1 year
Cecal intubation time | 1 year
Withdrawal time | 1 year
Polyps detection rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, China

IPD SHARING:
Plan to Share IPD: No